CLINICAL TRIAL: NCT01515488
Title: Assessing Utility of a "Kiosk Model" Self-Triage System in the Pediatric Emergency Department of A Tertiary Care Teaching Hospital
Brief Title: Kiosk-Model Self-Triage System in the Pediatric Emergency Department
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Valleywise Health (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2009-110; R03HS020235-01A1 (AHRQ)
Record Dates: First submitted 2012-01-13; First posted 2012-01-24 (Estimated); Results first posted 2012-10-15 (Estimated); Last update posted 2012-10-15 (Estimated); Status verified 2012-09

CONDITIONS: Emergencies
Keywords: Triage; Automated; Admitting; Pediatric ED
MeSH Terms: conditions — Emergencies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-triage kiosk (Experimental): Audio-assisted self-triage kiosk for obtaining medical history and presenting problem(s)
  Interventions: Other: Self-triage kiosk
- Nurse-initiated triage (Experimental): Nurse-initiated triage for obtaining medical history and presenting problem(s)
  Interventions: Other: Nurse-initiated triage

INTERVENTIONS:
Other: Nurse-initiated triage — Nurse-assisted triage for obtaining medical history and presenting problem(s)
  Other Names: standard triage
  Arms: Nurse-initiated triage
Other: Self-triage kiosk — Audio-assisted self-triage kiosk for obtaining medical history and presenting problem(s)
  Other Names: automated self-triage
  Arms: Self-triage kiosk

SUMMARY:
An audio-assisted self-triage kiosk in the Pediatric Emergency Department (ED) is expected to significantly reduce triage times, without any sacrifice of the quality of information that would be obtained by nurse-initiated triage.

DETAILED DESCRIPTION:
With the rapid evolution of consumer based information technology patients have the opportunity to become collaborative partners in their care. In addition, by bridging information gaps and improving workflow efficiency, continuity of care is optimized and the potential risk for error is reduced. Triage time for kiosk self-triage and nurse-initiated triage will be compared in terms of 1) triage time; 2) accuracy of medical history obtained; and 3) patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Between 0 and 18 years of age
* Registered in the Pediatric ED
* Accompanied by parent/guardian 18 years or older
* Version 3 Emergency Severity Index (ESI) of 3 to 5
* Parent or guardian able to communicate in English or Spanish

Exclusion Criteria:

* Deemed medically unstable
* ESI score of 1 or 2
* Incarcerated or in juvenile detention
* Parent/guardian unable to communicate in English or Spanish

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 400 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Madhumita Sinha, MD, MHSM, Principal Investigator — Valleywise Health
Locations (1):
- Maricopa Integrated Health System, Phoenix, Arizona, United States

REFERENCES:
- [Background] Morrison-Beedy D, Carey MP, Tu X. Accuracy of audio computer-assisted self-interviewing (ACASI) and self-administered questionnaires for the assessment of sexual behavior. AIDS Behav. 2006 Sep;10(5):541-52. doi: 10.1007/s10461-006-9081-y. PMID 16721506
- [Derived] Sinha M, Khor KN, Amresh A, Drachman D, Frechette A. The use of a kiosk-model bilingual self-triage system in the pediatric emergency department. Pediatr Emerg Care. 2014 Jan;30(1):63-8. doi: 10.1097/PEC.0000000000000037. PMID 24378865

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from the Pediatric Emergency Department at Maricopa Integrated Health System between February 2012 and April 2012.
Groups:
- Nurse-initiated Triage: Nurse-initiated triage for obtaining medical history and presenting problem(s)
  Nurse-initiated triage : Nurse-assisted triage for obtaining medical history and presenting problem(s)
- Self-triage Kiosk: Audio-assisted self-triage kiosk for obtaining medical history and presenting problem(s)
  Self-triage kiosk : Audio-assisted self-triage kiosk for obtaining medical history and presenting problem(s)
Period: Overall Study
Arm/Group | Nurse-initiated Triage | Self-triage Kiosk
Started | 200 | 200
Completed | 200 | 200
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Nurse-initiated Triage | Self-triage Kiosk | Total
Number analyzed (Participants) | 200 | 200 | 400
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 200 | 200 | 400
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 6 (6) | 6 (5) | 6 (5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 89 | 91 | 180
  Male | 111 | 109 | 220
Region of Enrollment [Number; unit: participants]
  United States | 200 | 200 | 400

OUTCOME MEASURES:

1. Primary Outcome: Triage Time
Description: The time it takes for the patient to be triaged, compared across the kiosk and nurse-initiated triage conditions.
Time Frame: From beginning of triage to completion of triage.
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | Nurse-initiated Triage | Self-triage Kiosk
Number analyzed (Participants) | 200 | 200
Seconds | 126.7 (62.6) | 94.4 (38.6)
Statistical Analysis 1: Comparison: Nurse-initiated Triage vs Self-triage Kiosk; Test type: Superiority or Other; p < 0.0005, t-test, 2 sided; DF=331.2; Mean Difference (Final Values) = 32.3, 95% CI 2-sided [22.1 to 42.6], Standard Error of Mean 5.2

2. Secondary Outcome: Accuracy of Medical History
Description: To check for accuracy of medical history information, two RAs approached enrolled parents during the course of their ED visit in the individual patient examination rooms. The RAs conducted a brief face-to-face interview with parents and verified information from the nursing triage summary sheet (for non-kiosk users) and the printout of history sheet from the kiosk users, noting any discrepancies on a Discrepancy Rating Scale. All historical discrepancies were categorized into three groups: major discrepancy, minor discrepancy and no discrepancy.
Time Frame: Upon completion of triage.
Measure: Mean (Standard Deviation); unit: Inaccuracies
Arm/Group | Nurse-initiated Triage | Self-triage Kiosk
Number analyzed (Participants) | 200 | 200
Inaccuracies | 1.03 (0.97) | 0.59 (0.81)

3. Secondary Outcome: Patient Satisfaction
Description: Custom survey with 4 items capturing satisfaction with Understanding, Ease of Answering Questions, Respect for Privacy, and Overall Feelings. For each item, the lowest possible score was 1 and the highest possible score was 6. For Understanding, the lowest actual score was 2 and the highest actual score was 6. For Ease of Answering Questions, the lowest actual score was 2 and the highest actual score was 6. For Respect for Privacy the lowest actual score was 3 and the highest actual score was 6. For Overall Feelings, the lowest actual score was 3 and the highest actual score was 6. For the (unweighted) average of all 4 items, the lowest possible score was 1 and the highest possible score was 6. The lowest actual score was 3.5 and the highest actual score was 6.0.
Time Frame: Upon completion of triage.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nurse-initiated Triage | Self-triage Kiosk
Number analyzed (Participants) | 200 | 200
units on a scale | 5.6 (0.8) | 5.7 (0.7)

ADVERSE EVENTS:
Description: No adverse events were possible; therefore no serious or other adverse events were reported.
Arm/Group | Nurse-initiated Triage | Self-triage Kiosk
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No